CLINICAL TRIAL: NCT03194152
Title: Effects of Peanut Consumption on Cardiovascular Disease Risk Factors and Gut Microbiota Among Adults in China: A Randomized Controlled Trial
Brief Title: Peanut Consumption and Cardiovascular Disease Risk in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Vasanti Malik, PI, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB17-0703
Record Dates: First submitted 2017-06-05; First posted 2017-06-21 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: T2D

STUDY DESIGN:
Intervention Model Description: Parallel design with two intervention arms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut (Experimental): Daily consumption of 2 servings of roasted peanuts for 12 weeks Intervention: Dietary Supplement: Roasted peanuts
  Interventions: Dietary Supplement: Peanut
- Control (Experimental): Daily consumption of isocaloric matched snack food for 12 weeks Intervention: Other: High Carbohydrate Snack
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Peanut — Dietary Supplement: Peanut
  Arms: Peanut
Dietary Supplement: Control — Dietary Supplement: High carbohydrate snacks
  Arms: Control

SUMMARY:
This is a 2 parallel-arm randomized controlled study with free-living subjects on self-selected diets. The objective of this study is to compare the effects of two servings of peanuts with an isocaloric matched refined carbohydrate snack food on glucose, lipids and lipoproteins and cardiovascular health risk factors, satiety and gut microbiota in 250 Chinese participants at risk for metabolic syndrome (overweight/obese, enlarged waist circumference, elevated LDL-cholesterol, prehypertension, and/or prediabetes).

The investigators hypothesize that the inclusion of 2 serving of peanuts in the diet will decrease blood glucose, LDL-cholesterol, and improve satiety sanctification between meals and gut microbiota compared to the control group and baseline.

DETAILED DESCRIPTION:
Emerging evidence has shown that peanut consumption has beneficial effects in modifying lipid profiles, glucose, and other cardiometabolic risk factors. During the last two decades, China has experienced a dramatic increase in T2D prevalence largely due to rapid social and economic growth. Peanuts are commonly consumed as snacks in China. However, there is limited evidence on the specific health benefits of peanuts as part of the Chinese habitual diet.

Clinical Study Protocol

Study diet Subjects will consume their habitual diet with the test snacks provided as roasted peanuts and rice flour snack bars twice a day during a mid- morning snack and mid -afternoon snack. Subjects in the peanut group will consume two serving of peanuts and subjects in the control group will consume isocaloric rice bars on a daily basis under on site supervision. Subjects will be instructed to maintain their habitual diet and physical activity. During the study period, body weight will be monitored routinely to ensure that baseline weight does not fluctuate by more than 1kg. Prior to day 1, day 42 and day 84, a three-day diet record will be administered to subjects to calculate basal energy intake.

Study design The study is a randomized, controlled, parallel-arm trial precedes by a 1-week run-in period with control treatment to assess compliance, acceptability and to determine baseline values.After the run-in period, participants will be randomized to either the control group or treatment group for three months. Each treatment phase will be 3 months in duration. At baseline, day 42 and day 84, clinical assessment (body weight, waist/hip circumference, blood pressure, pulse) will be preformed and blood samples will be collected. Urinary will be collected on baseline, day 42 and day 84. Fecal samples will be collected on baseline and day 84. Three days dietary records and appetite sensation ratings will be collected three times during the study (baseline, day 42 and day 84).

ELIGIBILITY:
Inclusion Criteria:

* 20-65
* Increased waist circumference : ≥ 90 cm for men and ≥ 80 cm for women

Plus 1 or more of the remaining criteria:

* Elevated TG level ≥ 1.7 mmo/L
* Reduced HDL-Cholesterol < 1.03 mmol/L in men and < 1.29 mmol/L in women)
* Fasting glucose ≥ 5.6 mmol/L
* Systolic/diastolic blood pressure ≥ 130/85 mmHg.

Exclusion Criteria:

* Taking lipid lowering medications
* With known or unknown peanut allergy (or any peanut containing products)
* Thyroid disease
* Diabetes mellitus
* Kidney disease
* Liver disease
* Cardiovascular disease or cancer
* Pregnant or lactating women
* Heavy alcohol consumption (>14 drinks/week)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Blood glucose will be measured at day 84.
  glucose, insulin, HbA1c

SECONDARY OUTCOMES:
Blood lipids level | Blood lipids level will be measured at day 84.
  cholesterol and triglyceride levels
Blood Inflammatory status | Inflammatory biomarkers will be measured at day 84.
  Inflammatory biomarkers
Assessment of appetite and other hunger sensations | Appetite and other hunger sensations will be measured at day 84.
  Appetite and other hunger sensations will be assessed using visual analogue scales
Microbiome | Micriobiome will be measured at day 84.
  fecal microbiome (subset) A subset of study subjects will be measured for fecal microbiome functionality.
Polyphenol metabolites | Polyphenol metabolites will be measured at day 84.
  Urinary polyphenol metabolites (subset)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoran Liu, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Liang Sun, Shanghai, China

REFERENCES:
- [Derived] Wang D, Sun L, Liu X, Niu Z, Chen S, Tang L, Zheng H, Chen X, Li H, Lu L, Malik V, Lin X. Replacing white rice bars with peanuts as snacks in the habitual diet improves metabolic syndrome risk among Chinese adults: a randomized controlled trial. Am J Clin Nutr. 2021 Jan 4;113(1):28-35. doi: 10.1093/ajcn/nqaa307. PMID 33236043